CLINICAL TRIAL: NCT05227612
Title: Psilocybin-assisted Cognitive Behavioral Therapy for Depression
Brief Title: Psilocybin-assisted CBT for Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Marc J. Weintraub, PhD, Assistant Clinical Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-002134; R34AT013077-01 (NIH)
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder
Keywords: psilocybin; cognitive behavioral therapy (CBT)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Psilocybin; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This study involves an open trial of 12 participant (i.e., all participants receive psilocybin-assisted cognitive behavioral therapy; PA-CBT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin + CBT (Experimental): Participants will receive 12 sessions of cognitive-behavioral therapy (CBT) along with two psilocybin-drug sessions -- the first following the third CBT session (10mg of psilocybin, taken orally) and the second following the sixth CBT session (25mg of psilocybin, taken orally).
  Interventions: Drug: Psilocybin; Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Drug: Psilocybin — Participants will receive two doses of psilocybin (10mg, 25mg).
Behavioral: Cognitive behavioral therapy — Twelve total sessions of therapy, including manualized cognitive behavioral therapy for major depressive disorder, including psychoeducation about depression, cognitive skills, and behavioral skills as well as preparation for psilocybin.

SUMMARY:
The primary objectives of this clinical investigation are to (1) determine the acceptability and feasibility of joining psilocybin-assisted therapy with cognitive-behavioral therapy (PA-CBT) for patients with depression, (2) optimize CBT to most effectively integrate the psilocybin experience with psychotherapy and (3) examine the clinical benefit of psilocybin as an adjunct to cognitive-behavioral therapy (CBT) for major depressive disorder.

This study will involve an open trial of PA-CBT where participants will receive two doses of psilocybin (10mg and then 25mg, separated by one month) plus 12 sessions of cognitive behavioral therapy.

ELIGIBILITY:
Inclusion Criteria:

* • Ages 21-60,

  * Able to swallow capsules,
  * Patients with a current major depressive episode or a history of major depressive episodes based on the DSM-5 criteria (American Psychiatric Association, 2013),
  * Active current depressive symptoms (i.e., scores >16 on the Hamilton-Depression Rating Scale (HAM-D) covering the prior 2 weeks; Hamilton, 1986),
  * Have an identified support person who can pick up the individual from UCLA Semel Institute and drive individual home following psilocybin sessions,
  * For women of child-bearing potential - using one form of highly effective contraception (e.g., oral contraceptive pill) and willingness to continue contraceptive use for duration of study
  * Patient has been medically cleared for the study by a physician.

Exclusion Criteria:

* • A personal or family history (first or second-degree) of psychosis or bipolar disorder

  * Resting blood pressure above 140 systolic, 90 diastolic (averaged across four separate measurements)
  * Meeting criteria for a DSM-5 cluster B personality disorder (narcissistic, histrionic, borderline, antisocial personality disorder),
  * Active suicidality (as indicated by a 3 or greater on item 3 of the HAM-D) or other psychiatric disturbance requiring acute treatment
  * Current use of antidepressants or other serotonergic-affecting substances (e.g., St. John's Wort and 5-hydroxytryptophan),
  * Currently receiving cognitive behavioral therapy,
  * Any of the following cardiovascular conditions: uncontrolled hypertension, coronary artery disease, congenital long QT syndrome, cardiac hypertrophy, cardiac ischemia, congestive heart failure, myocardial infarction, tachycardia, artificial heart valve, a clinically significant screening ECG abnormality, or any other significant cardiovascular condition
  * A history of stroke or Transient Ischemic Attack (TIA)
  * Epilepsy or history of seizures
  * Insulin-dependent diabetes
  * Meeting criteria for a DSM-5 substance abuse or dependence within prior 6 months
  * Positive urine drug screen for illicit substances
  * Use of other psychedelics or ketamine within prior 12 months
  * Adverse prior reaction to a psychedelic agent
  * Pregnant, trying to get pregnant, or nursing

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Treatment acceptability | 4-month treatment period
  participant and clinician feedback related to the joining of psilocybin with CBT
Treatment feasibility | 4-month treatment period
  recruitment and retention of participants in the trial
Hamilton Depression Rating Scale | 7-month study period
  symptom severity scored from 0-53, with larger values indicating greater depressive severity
Global Assessment of Functioning | 7-month study period
  psychosocial functioning scored from 0-100, with larger values indicating better functioning

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

REFERENCES:
- [Derived] Weintraub MJ, Jeffrey JK, Grob CS, Ichinose MC, Bergman RL, Cooper ZD, Miklowitz DJ. Psilocybin-Assisted Cognitive Behavioral Therapy for Adults with Major Depressive Disorder: Rationale and Treatment Development. Psychedelic Med (New Rochelle). 2023 Dec 13;1(4):230-240. doi: 10.1089/psymed.2023.0018. eCollection 2023 Dec. PMID 40046861